CLINICAL TRIAL: NCT05676151
Title: How Efficient is Music Therapy as a Distraction Technique in the Pain Rehabilitation Program Patients
Brief Title: Study of Music Therapy in Pain Rehabilitation Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher D. Sletten, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-003694
Record Dates: First submitted 2023-01-04; First posted 2023-01-09 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Music Therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy in Pain Rehabilitation (Experimental): Subjects undergoing care at the Mayo Clinic Florida Pain Rehabilitation Center (PRC) to address pain will receive a 20-minute music therapy intervention
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — 20-minute music-therapy-informed interventions (musical bingo, songwriting, lyric scramble) guided by a music therapist

SUMMARY:
The purpose of this study is to measure changes in mood, symptom burden, pain level, and stress scores in patients before and after a 20-minute music therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Patients that are enrolled in the Pain Rehabilitation Center, Mayo Florida

Exclusion Criteria:

- ≤ 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in mood | Baseline, after music intervention approximately 20 minutes
  We will use the NCCN distress thermometer before and after the creative work intervention to assess distress. For those patients who indicate high feelings of depression, their mood would be dealt with in accordance with clinic practice.
  The Distress Thermometer measures distress on a 0 to 10 scale. To report your distress, circle the number that matches your level of distress in the past week. The Problem List includes problems from 5 areas of life: practical, family, emotional, spiritual/religious, and physical problems. The higher the score the more distress experienced in that domain.
Change in pain level | Baseline, after music intervention approximately 20 minutes
  A 0-10 Likert Pain scale will be used. 0 = No Pain, 10 = Worst Pain Imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sletten, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials